CLINICAL TRIAL: NCT07285382
Title: A Multicenter, Randomized, Double-cohort Study of Different Doses of Dalpicicl Combined With Letrozole in the First-line Treatment of HR-positive, HER2-negative Advanced Breast Cancer
Brief Title: Different Doses of Dalpicicl Combined With Letrozole in the First-line Treatment of HR-positive, HER2-negative Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: wanghaibo (Other)
Responsible Party: Sponsor-Investigator, wanghaibo, PI, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dose optimization of dalpicicl
Record Dates: First submitted 2025-08-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: HR Positive HER2 Negative Advanced Breast Cancer
MeSH Terms: interventions — dalpiciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Dalpiciclib 125mg (Experimental): Participants receive dalpiciclib 125mg orally once daily plus letrozole 2.5mg orally once daily, continued until disease progression or unacceptable toxicity
  Interventions: Drug: Dalpiciclib 125mg; Drug: Letrozole 2.5mg
- Cohort B: Dalpiciclib 150mg (Experimental): Participants receive dalpiciclib 150mg orally once daily plus letrozole 2.5mg orally once daily, continued until disease progression or unacceptable toxicity
  Interventions: Drug: Dalpiciclib 150mg; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Dalpiciclib 125mg — Oral administration, 125mg，Dalpiciclib is administered for 3 weeks, followed by 1 week of rest
  Arms: Cohort A: Dalpiciclib 125mg
Drug: Dalpiciclib 150mg — Oral administration, 150mg，Dalpiciclib is administered for 3 weeks, followed by 1 week of rest
  Arms: Cohort B: Dalpiciclib 150mg
Drug: Letrozole 2.5mg — Oral administration, 2.5mg, administered once daily until disease progression or unacceptable toxicity

SUMMARY:
This study is a prospective, open-label, randomized, multicenter, two-cohort phase II clinical trial. Starting from December 1, 2024, it plans to enroll 120 patients with advanced first-line HR-positive, HER2-negative breast cancer. A centralized randomization system (IWRS) will be used for randomization, and stratification will be performed based on the following factors during randomization: 1) Visceral metastasis (yes vs no); 2) Disease-free interval (previously untreated vs 12 < DFI ≤ 24 vs DFI > 24).

Cohort A: Dalpiciclib 125mg + Letrozole 2.5mg Cohort B: Dalpiciclib 150mg + Letrozole 2.5mg Imaging assessment will be conducted in accordance with the RECIST 1.1 criteria, and tumor imaging evaluation will be performed by investigators from the participating centers.

Patients receiving dalpiciclib will undergo a safety visit 28 days after the last dose, followed by survival follow-up until the patient's death or trial termination (whichever comes first).

Pharmacokinetic assessment: Blood samples will be collected once before dosing on Cycle 1 Day 15 (C1D15), 4 hours after dosing on C1D15, before dosing on Cycle 2 Day 1 (C2D1), and before dosing on Cycle 4 Day 1 (C4D1) to explore the population pharmacokinetic characteristics of dalpiciclib and the factors affecting its pharmacokinetics. The first dosing time of the subjects, each blood collection time, the dalpiciclib dosing time within three days before blood collection, and the dalpiciclib dosing time on the day of C1D15 blood collection must be accurately recorded. If dalpiciclib is not administered within 14 days before the planned PK blood collection, no PK blood collection will be performed on the day of that visit. If possible, PK samples should be collected simultaneously with samples for other laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years and ≤75 years, who are postmenopausal or premenopausal/perimenopausal, and meet one of the following conditions:

  1. Have undergone bilateral oophorectomy in the past, or be aged ≥60 years; or
  2. Aged <60 years, in a natural postmenopausal state (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), with E2 and FSH at postmenopausal levels; or
  3. Premenopausal or perimenopausal female patients can also be enrolled, but must be willing to receive LHRH agonist treatment during the study period
* Patients with breast cancer confirmed by pathological examination to be HR-positive and HER2-negative, with evidence of focal recurrence or metastasis, not suitable for surgical resection or radiotherapy with the goal of cure, and without clinical indications for chemotherapy.

  1. ER-positive and/or PR-positive is defined as: the proportion of tumor cells with positive staining among all tumor cells is ≥1% (reviewed and confirmed by the investigator at the participating trial center);
  2. HER2-negative is defined as: standard immunohistochemistry (IHC) test result is 0/1+; ISH test shows that the HER2/CEP17 ratio is less than 2.0 or the HER2 gene copy number is less than 4 (reviewed and confirmed by the investigator at the participating trial center)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1
* Have not previously received any systemic antineoplastic treatment for focal recurrent or metastatic disease
* Have measurable lesions in line with RECIST 1.1 criteria or only bone metastatic lesions (including osteolytic lesions or mixed osteolytic/osteoblastic lesions)
* Have sufficient organ and bone marrow function
* Women of childbearing potential must be willing to use a medically approved highly effective contraceptive method during the study period and within 3 months after the last administration of the study drug
* All acute toxic effects of previous antineoplastic treatment have resolved to grade 0-1 (according to NCI-CTCAE Version 5.0) or to the level specified in the inclusion/exclusion criteria. Except for other toxicities such as alopecia that the investigator deems to pose no safety risk to the patient
* Have given informed consent and signed the informed consent form, and be willing and able to comply with the planned visits, study treatment plan, laboratory tests and other trial procedures

Exclusion Criteria:

* Previously diagnosed with HER2-positive breast cancer by pathological examination
* Inflammatory breast cancer
* Disease progression or recurrence at 12 months or within 12 months after completion of previous neoadjuvant or adjuvant endocrine drug treatment
* Patients judged by the investigator to be unsuitable for endocrine treatment. Including advanced patients with symptoms, disseminated to internal organs, and at risk of life-threatening complications in the short term (including those with uncontrollable large effusions [pleural, pericardial, peritoneal], lymphangitis of the lung, and patients with more than 50% liver involvement) Confirmed to have brain metastatic lesions by cranial CT or MRI examination
* Have previously received any CDK4/6 inhibitor drug treatment
* Underwent major surgery, chemotherapy, radiotherapy, any investigational drug or other anticancer treatment within 2 weeks before entering the study Diagnosed with any other malignant tumor within 3 years before entering the study, except for non-melanoma skin cancer, basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix that have undergone radical treatment Human Immunodeficiency Virus (HIV) infection or known to have Acquired Immunodeficiency Syndrome (AIDS), active hepatitis B (HBV DNA ≥1000 IU/ml), hepatitis C (positive hepatitis C antibody and HCV-RNA higher than the lower limit of detection of the analytical method), or co-infection with hepatitis B and hepatitis C
* Within 6 months before entering the study, the following occurred: myocardial infarction, severe/unstable angina pectoris, NYHA class 2 or higher cardiac insufficiency, persistent arrhythmia of grade ≥2 (according to NCI-CTCAE Version 5.0), atrial fibrillation of any grade, coronary/peripheral artery bypass surgery, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism)
* Complicated with severe infection within 4 weeks before the first administration (e.g., requiring intravenous infusion of antibiotics, antifungal or antiviral drugs according to clinical diagnosis and treatment norms), or unexplained fever >38.5℃ during the screening period/before the first administration
* Inability to swallow, intestinal obstruction, or other factors that affect drug administration and absorption
* Known allergy to the study drug or any excipients
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Known history of psychiatric drug abuse or drug addiction
* Patients currently participating in other studies
* Have other serious physical or mental diseases or laboratory test abnormalities that may increase the risk of participating in the study, interfere with the study results, and are deemed unsuitable for participating in this study by the investigator

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression - Free Survival (PFS) | From date of randomization until the date of first documented disease progression or death from any cause (whichever comes first), assessed per RECIST 1.1 criteria up to 104 weeks
  Progression - Free Survival (PFS) is registered as 'Primary' as the most clinically impactful endpoint; other outcomes (ORR, DoR) are secondary per platform requirements, though protocol does not hierarchy
Duration of Response (DoR) | From the date of first documented complete response (CR) or partial response (PR) (per RECIST 1.1, assessed by investigators via imaging) until the date of first documented disease progression (per RECIST 1.1) or recurrence, assessed up to 104 weeks
  Time from first documentation of complete response (CR) or partial response (PR) to disease progression (per RECIST 1.1) or recurrence, assessed by investigators via imaging

OTHER OUTCOMES:
Objective Response Rate, ORR | From date of randomization until the date of first documented disease progression or trial completion (whichever comes first), assessed per RECIST 1.1 criteria up to 104 weeks
  Proportion of participants with complete response (CR, disappearance of all target lesions) or partial response (PR, ≥ 30% reduction in sum of target lesion diameters) per RECIST 1.1.
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 208 weeks (4 years)
  Time from randomization to death from any cause, with survival status monitored until trial completion or participant withdrawal.
Patient - Reported Outcome (PRO): Quality of Life | From baseline, then every 3 weeks during study treatment, until the date of trial completion (assessed up to 104 weeks)]
  Quality of life assessed via EORTC QLQ - C30 questionnaire (score range: 0-100; for functional domains, higher scores indicate better quality of life; for symptom domains, higher scores indicate more severe symptoms), focusing on physical, emotional, and functional well - being. Administered at baseline, then every 3 weeks during treatment until trial completion.
Safety: Adverse Event Profile | From first dose until 30 days after last dose, monitored continuously
  Adverse events (AEs) assessed by CTCAE v5.0 criteria, including type, severity, and duration. Monitored from first dose until 30 days after last dose

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Qingdao University Affiliated Hospital, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: Undecided